CLINICAL TRIAL: NCT03872986
Title: Clinical Evaluation of Caries Sealing Technique on Primary Teeth Using Giomer and Glass Ionomer Cement (GIC) With or Without Silver Diamine Fluoride (SDF)
Brief Title: Caries Sealing Using Giomer and Glass Ionomer Cement With or Without Silver Diamine Fluoride
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Caries sealing
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Caries, Dental; Caries Class I
Keywords: primary teeth; silver diamine fluoride; caries sealing
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SDF+Giomer (Experimental): Combined Silver Diamine Fluoride (SDF) and Potassium Iodide (KI) + Beautifil II restorative material
  Interventions: Device: SDF; Device: Giomer
- Giomer only (Experimental): Beautifil II dental restorative material
  Interventions: Device: Giomer
- SDF+GIC (Experimental): Combined Silver Diamine Fluoride (SDF) and Potassium Iodide (KI) + Equia forte
  Interventions: Device: SDF; Device: GIC
- GIC only (Experimental): Equia forte dental restorative material
  Interventions: Device: GIC

INTERVENTIONS:
Device: SDF — Combined Silver Diamine Fluoride (SDF) and Potassium Iodide (KI)
  Arms: SDF+GIC; SDF+Giomer
Device: Giomer — Beautifil II dental restorative material
  Arms: Giomer only; SDF+Giomer
Device: GIC — Equia forte dental restorative material
  Arms: GIC only; SDF+GIC

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of Giomer and GIC restorations with and without SDF on caries sealing of primary molar teeth

DETAILED DESCRIPTION:
Restorations will be placed on four primary molar teeth with occlusal caries, in a split mouth design. 100 patients will be included in the study. The teeth will be randomized into four groups according to the restorative materials.

Group 1: SDF (Riva Star) + Giomer (Beautifil II, (Shofu Dental, Tokyo, Japan) Group 2: Giomer (Beautifil II, (Shofu Dental, Tokyo, Japan) Group 3: SDF (Riva Star) + GIC (Equia Forte, GC, Japan) Group 4: GIC (Equia Forte, GC, Japan)

The restorations will be evaluated clinically at baseline and 6., 12., 18., 24. months and radiologically at 6., 12. and 24. months. The modified US Public Health Service criteria (secondary caries, marginal integrity, marginal discoloration and retention) will be used for clinical evaluation of restorations. Intra-oral photos will be taken directly after treatment and at control appointments.

The data will be analysed statistically using Wilcoxon test, chi square test and the Kaplan-Meier survival method will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of the patients who accept to participate and sign the informed consent.
* Patients who have at least four first and/or second primary molars that require class I restorations
* Teeth that have healthy lamina dura and periodontal ligament
* Teeth that have caries lesions not extending to the pulp radiographically
* Patients whose first molar teeth are in occlusion

Exclusion Criteria:

* Patients and parents of the patients who does not accept to participate and sign the informed consent
* Teeth which need endodontic treatment
* Teeth that have caries more than one surface
* Teeth that are previously restored
* Patients who are not cooperative for the dental procedure
* Teeth that doesn't have proximal or occlusal contacts with adjacent healthy teeth
* Patients who have bruxism, skeletal or dental malocclusion
* Teeth that have developmental defects/anomalies or discoloration
* Patients who have allergies to resin based restorative materials

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The US Public Health Service criteria for secondary caries on restorations | 2 years
  A:There is no clinical diagnosis of caries C:There is clinical diagnosis of caries
The US Public Health Service criteria for retention of restorations | 2 years
  Alpha: No loss on the restoration Bravo:Partial loss on the restoration Charlie:Total loss on the restoration
The US Public Health Service criteria for marginal discoloration on restorations | 2 years
  Alpha: No visual evidence of discoloration Bravo: Slight staining which can be polished away Charlie: Discoloration has penetrated in the pulpal direction
The US Public Health Service criteria for marginal adaptation on restorations | 2 years
  Alpha: Restoration is fully intact. No explorer catch evident Bravo: Slight explorer catch in no more than 1/3 of margins Charlie: Explorer catch and/or penetration is evident in more than 1/3 of restoration margin
The US Public Health Service criteria for surface roughness on restorations | 2 years
  Alfa: Enamel-like surface Bravo: Surface rougher than enamel, clinically acceptable Charlie: Surface unacceptably rough / restoration is broken or cracked
The US Public Health Service criteria for anatomical form on restorations | 2 years
  A: No loss on anatomical form of the restoration B: Change in anatomical form but dentin or cement is not expose C: Change in anatomical form that expose dentin or cement

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Cehreli, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara
  - Hacettepe university, Ankara

IPD SHARING:
Plan to Share IPD: Undecided